CLINICAL TRIAL: NCT00734214
Title: Hypotonic Versus Isotonic Parenteral Fluids in Children - a Randomized Controlled Trial
Brief Title: Hypotonic Versus Isotonic Parenteral (HIP) Fluid Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-265
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2012-06-13 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hyponatremia; Hypernatremia
Keywords: Parenteral Fluids; Isotonic; Hypotonic; Pediatric; Fluid overload
MeSH Terms: conditions — Hyponatremia; Hypernatremia; Edema | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.9% NaCl (Experimental)
  Interventions: Drug: 0.9% NaCl
- 0.45% NaCl (Active Comparator)
  Interventions: Drug: 0.45%NaCl

INTERVENTIONS:
Drug: 0.9% NaCl — Intravenous Fluid
  Isotonic Parenteral Fluid
  Other Names: Isotonic saline
  Arms: 0.9% NaCl
Drug: 0.45%NaCl — Intravenous Fluid
  Hypotonic Parenteral Fluid
  Other Names: Hypotonic saline
  Arms: 0.45% NaCl

SUMMARY:
Children who are undergoing surgery need intravenous fluids to prevent dehydration and maintain their electrolyte balance. The current standard of care in these children is to use a fluid which is low in sodium (hypotonic fluid). The safety of this practice has never been tested. There is ongoing concern from the medical community that this type of fluid increases the child's risk of developing low sodium levels, and hence may not be safe for all children. Low sodium can lead to significant complications such as seizures, coma and even death, risks of which are often underestimated and not anticipated by their caregivers. Experts in the field suggest that giving a solution with a similar sodium content to that of blood (isotonic fluid) reduces the risk of these problems in these children. This study will compare these two types of intravenous fluids (hypotonic versus isotonic), in a blinded fashion (i.e. neither the patient nor caregivers or investigators will be aware which type of fluid the patient is receiving), in children following surgery. The investigators goal is to see which type of fluid is safer, and leads to more stable sodium levels. This would in turn lead to a lower risk of complications as described above.

This is the first time such a study is preformed in pediatrics. There are unnecessary number of complications and potential deaths from this disorder, and hence the safety of everyday fluid practice in children needs to be scientifically tested. The results of this study will enable the investigators to propose scientifically based guidelines on how to minimize risks associated with intravenous infusions in children.

DETAILED DESCRIPTION:
Research Question:

In general pediatric surgical patients, do isotonic PMS compared to hypotonic PMS, result in a lower risk of acute hospital acquired plasma sodium derangements, occurring at any time during the study intervention? Primary efficacy objective -To determine the impact of postoperative administration of isotonic compared to hypotonic PMS on the risk of hospital acquired PNa derangements in pediatric surgical patients, occurring at any time during the study intervention.

Secondary efficacy objectives: a) To determine the impact of postoperative administration of isotonic compared to hypotonic PMS on clinical sequelae related to acute PNa changes, in pediatric surgical patients. b) the independent predictors of hospital acquired PNa derangements will be explored.

Study Design:

This is a double-blind randomized controlled trial. Participants, health care providers, data collectors, and judicial assessors of outcomes will be blinded to the study intervention.

Setting: McMaster Children's Hospital.

Trial Intervention:

Enrolled patients will be randomized postoperatively to receive either one of the following parenteral maintenance solutions: 1) hypotonic PMS, or 2) isotonic PMS. For the purposes of this study the hypotonic PMS will be 0.45%NaCl, and the Isotonic PMS will be 0.9% NaCl. Enrolled patients will receive their allocated treatment (provided there are no safety issues or concerns) until they are fully orally fed and the PMS rate is no greater than a rate required to "keep vein open (KVO)", to a maximum duration of 48 hours. The physician can thereafter administer the maintenance solution of their choice. The following parameters will be monitored in each study participant during the treatment period: hourly urine output, strict intake and output, 12 hourly fluid balances and daily weights. Blood and urine samples will be obtained on study patients every 12 hours until they are fully orally fed and the IV rate is at KVO, for a maximum of 48 hours. Any additional investigations ordered by the caring physician during the treatment and follow up period will also be recorded. Patients will be followed for clinical outcomes for 48 hours after the study intervention is discontinued, or until the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, 6 months corrected age -16 years, undergoing surgery.
* Within 6 hours of the immediate post-operative period.
* Post-operative stay anticipated to be more than 24 hours.
* Primary route of fluid administration is anticipated to be intravenous, in the first 24 hours following surgery.
* Informed consent of parent/guardian.
* Consent to participate from surgeon.

Exclusion Criteria:

* Patients under 6 months of age
* Patients equal to or over 17 years of age
* Patients with hemodynamic instability , defined as a requirement for continuous vasoactive infusion (e.g. epinephrine, dopamine, norepinephrine, phenylephrine, milrinone, or Dobutamine) to maintain blood pressure at the end of surgery.
* Patients admitted into the "short stay" post-operative unit
* Patients in whom either hypotonic or isotonic solutions may be contraindicated/necessary: i.e. specific neurosurgical patients (ie those at risk of increased ICP, e.g. requiring actual brain surgery, ICP monitor or external ventricular drain insertion), patients with diabetic ketoacidosis, acute (≤ 7 days) burns, pre-existing CHF, liver failure or cirrhosis, renal failure.
* Patients with known pre-existing risk of PNa derangements: DI or SIADH
* Chronic diuretic use - defined as use of any oral or intravenous diuretics for ≥ 7 days.
* Known, uncorrected PNa derangement (PNa < 134 or > 146 mmol/L), identified peri-operatively (i.e. within 12 hours of surgery or during surgery).
* Prior enrolment in this study
* Patients or their guardians objecting to give consent.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MB, BCh, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Choong K, Arora S, Cheng J, Farrokhyar F, Reddy D, Thabane L, Walton JM. Hypotonic versus isotonic maintenance fluids after surgery for children: a randomized controlled trial. Pediatrics. 2011 Nov;128(5):857-66. doi: 10.1542/peds.2011-0415. Epub 2011 Oct 17. PMID 22007013

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.9% NaCl | 0.45% NaCl
Started | 128 | 130
Completed | 124 | 126
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 4
Not completed — MD withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.9% NaCl | 0.45% NaCl | Total
Number analyzed (Participants) | 128 | 130 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 128 | 130 | 258
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (5.5) | 9.2 (5.7) | 9.2 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 68 | 143
  Male | 53 | 62 | 115
Region of Enrollment [Number; unit: participants]
  Canada | 128 | 130 | 258

OUTCOME MEASURES:

1. Primary Outcome: Hospital Acquired Acute Plasma Sodium Derangements (Hypo- or Hypernatremia)
Time Frame: During the treatment and follow-up period.
Reporting Status: Not Posted

2. Secondary Outcome: Adjudicated Morbidity Attributed to Acute Plasma Sodium Changes.
Time Frame: During the treatment and follow-up period
Reporting Status: Not Posted

3. Primary Outcome: Hyponatremia
Description: Plasma sodium less than 135 mmol/L
Time Frame: during the study intervention
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | 0.9% NaCl | 0.45% NaCl
Number analyzed (Participants) | 128 | 130
participants | 29 | 53

ADVERSE EVENTS:
Arm/Group | 0.9% NaCl | 0.45% NaCl
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/130
Other Adverse Events (participants affected / at risk) | 9/128 | 8/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.9% NaCl (N=128) | 0.45% NaCl (N=130)
Generalized edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
New onset hypertension (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.9% NaCl (N=128) | 0.45% NaCl (N=130)
Generalized Edema (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (10)
New onset Hypertension (Blood and lymphatic system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No